CLINICAL TRIAL: NCT02109965
Title: The Effect of Dexmedetomidine on the Microcirculation in Patients With Severe Sepsis and Septic Shock
Brief Title: The Effect of Dexmedetomidine on Microcirculation in Severe Sepsis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201311031MINB
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — Dexmedetomidine; Midazolam; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Use midazolam or propofol for sedation
  Interventions: Drug: Midazolam; Drug: Propofol
- Dexmedetomidine (Experimental): Use dexmedetomidine for sedation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Continue infusion (CIF) 0.1 - 0.7 mcg/kg/h Goal of sedation: Richmonad agitation-sedation scale 0 to -2
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Midazolam — CIF Goal of sedation: Richmonad agitation-sedation scale 0 to -2
  Other Names: Dormicium
  Arms: Control
Drug: Propofol — CIF Goal of sedation: Richmonad agitation-sedation scale 0 to -2
  Other Names: Propofol-Lipuro
  Arms: Control

SUMMARY:
Despite early goal-directed maintenance of normal macrocirculation, the reduction of 60-day mortality of patients with severe sepsis and septic shock remained unsatisfied (56.9% to 44.3%). One of the major causes of high mortality is microcirculatory dysfunction. Delayed diagnosis and treatment of microcirculatory dysfunction may cause tissue hypoperfusion and resulted in multiple organ dysfunction and death. Dexmedetomidine is a highly selective α2-adrenoreceptor agonist which exhibits sedative and analgesic effects. Recent studies suggest that dexmedetomidine also has anti-coagulation and anti-inflammatory effects, and it can reduce the mortality of endotoxemic rats and patients with severe sepsis. The investigators will conduct two animal studies and one clinical trial to investigate the effect of dexmedetomidine on microcirculatory dysfunction and organ injury in rat with endotoxemia and patients with severe sepsis and septic shock.

Sixty patients with severe sepsis and septic shock will be enrolled and randomized to control group or dexmedetomidine group. In the control group, the patients will be treated according to the clinical practice guideline. If sedation is required, non-dexmedetomidine sedative agents will be used. In the dexmedetomidine group, the patients will be treated according to the clinical practice guideline, and they will also receive continuous infusion of dexmedetomidine (infusion rate ranged from 0.1 to 0.7 mcg/kg/h) for 24 hours as needed. The sublingual microcirculation, serum level of Endocan, NGAL(Neutrophil Gelatinase-Associated Lipocalin), and BNP(B-type natriuretic peptide) will be examined at preset time points up to 24 hours. The vital signs, hemodynamic parameters, and survival of 28-day and 90-day will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients who require sedation
* Patients who have diagnosis of severe sepsis / septic shock
* meet 2 or more of the 4 SIRS criteria
* with one organ dysfunction according the definition of Surviving Sepsis Campaign

Exclusion Criteria:

* less than 20 y/o
* refractory bradycardia (heart rate slower than 60 bpm despite of adequate treatment)
* 2nd and 3rd degree of AV-block
* the onset of severe sepsis/septic shock is more than 24h before enrollment
* APACHE II > 30 at enrollment
* Severe liver cirrhosis (Child B or C)
* New onset of myocardial infarction within 30 days or heart failure (NYHA 4)
* attend other trial in ICU within one month
* patient who is pregnant
* receive organ transplantation within one year
* expected survival is less than 30 days by attending physician
* receive cardiopulmonary resuscitation within 4 weeks
* patients who have signed consent of refusal of cardiopulmonary resuscitation and invasive therapy
* have allergic history to dexmedetomidine
* receive renal replacement therapy within 24 hours before enrollment
* patient with HIV infection
* non-native speaker
* other factors not eligible for enrollment concerned by attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02-24 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Changes of total small vessel density and perfused small vessel density | 6h

SECONDARY OUTCOMES:
Changes of total small vessel density and perfused small vessel density | 24h
Change of microvascular flow index | 6h and 24h

OTHER OUTCOMES:
Endocan level | 24h
Hemodynamic variables | 6h and 24h
  Use EV1000 clinical platform MAP HR Cardiac index Stroke volume index Systemic vascular resistance index
NGAL level | 6h and 24h
  Neutrophil Gelatinase-Associated Lipocalin
BNP level | 24h
  B-type natriuretic peptide)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan